CLINICAL TRIAL: NCT05406323
Title: The Effect of Web - Based Fall Prevention Program on Fall, Fall Risk and Fall Fear Among Elderly
Brief Title: Web-Based Fall Prevention Program for Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nur Sema KAYNAR, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IUC-YYU
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Fall; Fall Risk; Fear of Falling
Keywords: fall prevention; web-based intervention; elderly; Falling; Fear of Falling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Fall Prevention Program Intervention (Experimental): Participants in this group will receive a 6-week Web-Based Fall Prevention Program intervention, comprising of health education, exercise and safe home environment. Web-Based Fall Prevention Program will be conducted on web based (Web - Based Fall Prevention Program website)
  Interventions: Behavioral: Web-Based Fall Prevention Program
- Control Group (No Intervention): The control group will not receive any intervention during the study. Participants in the control group will take the same program after the study is complete.

INTERVENTIONS:
Behavioral: Web-Based Fall Prevention Program — Health education: This intervention consisted of seven health issues which are "Fall among elderly", "fall risk factors", " fall prevention interventions-exercise", " fall prevention interventions-healthy diet", " fall prevention interventions- drug use", "fall prevention interventions- vision", "fear of falling".
  Exercise: This intervention is the exercise that is a combination of balance and strengthening exercises (8 exercise). Participants will do the exercises at least three days a week (along 6 week).
  Safe home environment: This intervention is aimed at providing a fall-safe home environment for the participants. In this context, the participants will watch the video on creating a safe home environment for falling. Participants will also be asked to answer the "Home Safety Check Form for Falls" to make their home more fall-proof. In this form, according to the answers given by the participants, suggestions will be given to prevent the risks of falling in the home environment.
  Arms: Web-Based Fall Prevention Program Intervention

SUMMARY:
Fall is one of the most common problems experienced by the elderly, is an important public health problem in many societies. Falls are one of the leading causes of fatal and non-fatal injuries in the elderly. An average of one-third of individuals aged 65 and over have a fall at least once each year. The research will be carried out on the web page that on fall prevention prepared within the scope of this project. The aim of this project is to assess the effect of Web-Based Fall Prevention Program on falling, fall risk and fear of fall.

DETAILED DESCRIPTION:
The research was planned as a experimental design with a pretest- posttest control group design. It will be with individuals over the age of 65. The sample size of the research is consists of 72 people who agreed to participate in the research. Participant will be randomly assigned to the experimental and control groups via computer programı (random.org).

The research will be conduct on a web-based basis.The six-week web-based program includes health education, exercise and safe home environment initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study,
* 65 years or older,
* Completing the Timed Up and Go (TUG) test for 12 seconds or more,
* Having internet access and the ability to use communication tools such as computers, tablets or smartphones,
* Not dependent on bed,
* Without moderate and severe cognitive impairment (Mini Mental State Test-MMD ≥24),

Exclusion Criteria:

* Illiterate,
* Visually impaired,
* Physical condition or disease that may prevent exercise (Multiple Sclerosis, Parkinson, with a fracture, artificial knee- hip-joint in the last six months etc..)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Change in number of falls | Pre, post (6 weeks), 3 months, 6 months
  Participants will be asked about the number of falls in the past 12 months
Change in Fall Risk | Pre, post (6 weeks), 3 months, 6 months
  Simple screening test that is a sensitive and specific measure of probability for falls among older adults. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.
Change in Falls Efficacy Scale (FES) | Pre, post (6 weeks), 3 months, 6 months
  Falls Efficacy Scale (FES) was developed to assess individuals' fear of falling. It consists of 10 items. The items are answered with yes or no. An increase in the individual's fear of falling mean score means that the fear of falling increases.

SECONDARY OUTCOMES:
Change in The Falls Behavioral (FaB) Scale | Pre, post (6 weeks), 3 months, 6 months
  It has 30 items and 10 dimensions, and it is designed to identify an older person's awareness of-and practice of-behaviors that could potentially protect the individual from falling. The 10 behavioral dimensions were cognitive adaptations, protective mobility, avoidance, awareness, pace, practical strategies, displacing activities, being observant, changes in level, and getting to the phone. Items of the scale are based on self-reporting and were scored from 1 (never) to 4 (always), with 0 for does not apply. Increases in subscales' mean scores indicate the individual is making safe behavioral changes or not taking risky behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Sema KAYNAR, MSc, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No